CLINICAL TRIAL: NCT01204684
Title: A Phase II Clinical Trial Evaluating Autologous Dendritic Cells Pulsed With Tumor Lysate Antigen +/- Toll-like Receptor Agonists for the Treatment of Malignant Glioma
Brief Title: Dendritic Cell Vaccine for Patients With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-000202
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Glioma; Anaplastic Astrocytoma; Anaplastic Astro-oligodendroglioma; Glioblastoma
Keywords: dendritic cells; glioma; vaccine; glioma of WHO Grade III or IV
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tumor Lysate-pulsed DC vaccination (Experimental): Cohort #1 will receive autologous tumor lysate-pulsed DC vaccination together with a placebo cream or intramuscular injection of saline.
  Interventions: Biological: autologous tumor lysate-pulsed DC vaccination
- Tumor lysate-pulsed DC vaccination+0.2% resiquimod. (Experimental): Cohort #2 will receive autologous tumor lysate-pulsed DC vaccination together with adjuvant 0.2% resiquimod.
  Interventions: Biological: Tumor lysate-pulsed DC vaccination+0.2% resiquimod
- Tumor-lysate pulsed DC vaccination +adjuvant polyICLC. (Experimental): Cohort #3 will receive autologous tumor lysate-pulsed DC vaccination together with adjuvant poly ICLC (TLR3 agonist).
  Interventions: Biological: Tumor-lysate pulsed DC vaccination +adjuvant polyICLC

INTERVENTIONS:
Biological: autologous tumor lysate-pulsed DC vaccination
  Arms: Tumor Lysate-pulsed DC vaccination
Biological: Tumor lysate-pulsed DC vaccination+0.2% resiquimod
  Arms: Tumor lysate-pulsed DC vaccination+0.2% resiquimod.
Biological: Tumor-lysate pulsed DC vaccination +adjuvant polyICLC
  Arms: Tumor-lysate pulsed DC vaccination +adjuvant polyICLC.

SUMMARY:
The main purpose of this study is to evaluate the most effective immunotherapy vaccine components in patients with malignant glioma. Teh investigators previous phase I study (IRB #03-04-053) already confirmed that this vaccine procedure is safe in patients with malignant brain tumors, and with an indication of extended survival in several patients. However, the previous trial design did not allow us to test which formulation of the vaccine was the most effective. This phase II study will attempt to dissect out which components are most effective together. Dendritic cells (DC) (cells which "present" or "show" cell identifiers to the immune system) isolated from the subject's own blood will be treated with tumor-cell lysate isolated from tumor tissue taken from the same subject during surgery. This pulsing (combining) of antigen-presenting and tumor lysate will be done to try to stimulate the immune system to recognize and destroy the patient's intracranial brain tumor. These pulsed DCs will then be injected back into the patient intradermally as a vaccine. The investigators will also utilize adjuvant imiquimod or poly ICLC (interstitial Cajal-like cell) in some treatment cohorts. It is thought that the host immune system might be taught to "recognize" the malignant brain tumor cells as "foreign" to the body by effectively presenting unique tumor antigens to the host immune cells (T-cells) in vivo.

ELIGIBILITY:
PATIENT ELIGIBILITY

Inclusion Criteria

1. Patients with newly diagnosed or recurrent glioma of WHO Grade III or IV {anaplastic astrocytoma (AA), anaplastic astro-oligodendroglioma (AO), or glioblastoma (GBM)} will be eligible for this protocol.
2. Patients must have had surgical resection at UCLA (University of California, Los Angeles), for which a separate informed consent was signed for the collection of their tumor prior to surgery.
3. After surgery, a pathological diagnosis of malignant glioma (WHO Grade III or IV) will need to be established.
4. Patients must be 18 years or older and able to read and understand the informed consent document. Patients must sign the informed consent indicating that they are aware of the investigational nature of this study.
5. Patients must have a Karnofsky performance status (KPS) rating of > 60 prior to initiating treatment. Patients may be enrolled at a KPS of < 60 if it is felt that the patient will have adequate opportunity to recover to a KPS of > 60 by the initiation of treatment.

Exclusion Criteria

1. Subjects with an active infection.
2. Inability to obtain informed consent because of psychiatric or complicating medical problems.
3. Unstable or severe intercurrent medical or psychiatric conditions as determined by the Investigator.
4. Females of child-bearing potential who are pregnant or lactating or who are not using approved contraception.
5. History of immunodeficiency (e.g., HIV) or autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, vasculitis, polymyositis-dermatomyositis, scleroderma, multiple sclerosis, or juvenile-onset insulin-dependent diabetes) that may be exacerbated by immunotherapy.
6. Subjects with organ allografts.
7. Inability or unwillingness to return for required visits and follow-up exams.
8. Subjects who have an uncontrolled systemic malignancy that is not in remission.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Most effective combination of DC vaccine components | 6 weeks

SECONDARY OUTCOMES:
Time to tumor progression and overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Los Angeles, California, Los Angeles, California, United States

REFERENCES:
- [Background] Liau LM, Black KL, Prins RM, Sykes SN, DiPatre PL, Cloughesy TF, Becker DP, Bronstein JM. Treatment of intracranial gliomas with bone marrow-derived dendritic cells pulsed with tumor antigens. J Neurosurg. 1999 Jun;90(6):1115-24. doi: 10.3171/jns.1999.90.6.1115. PMID 10350260
- [Background] Liau LM, Prins RM, Kiertscher SM, Odesa SK, Kremen TJ, Giovannone AJ, Lin JW, Chute DJ, Mischel PS, Cloughesy TF, Roth MD. Dendritic cell vaccination in glioblastoma patients induces systemic and intracranial T-cell responses modulated by the local central nervous system tumor microenvironment. Clin Cancer Res. 2005 Aug 1;11(15):5515-25. doi: 10.1158/1078-0432.CCR-05-0464. PMID 16061868
- [Background] Prins RM, Liau LM. Cellular immunity and immunotherapy of brain tumors. Front Biosci. 2004 Sep 1;9:3124-36. doi: 10.2741/1465. PMID 15353342
- [Background] Prins RM, Cloughesy TF, Liau LM. Cytomegalovirus immunity after vaccination with autologous glioblastoma lysate. N Engl J Med. 2008 Jul 31;359(5):539-41. doi: 10.1056/NEJMc0804818. No abstract available. PMID 18669440
- [Derived] Everson RG, Hugo W, Sun L, Antonios J, Lee A, Ding L, Bu M, Khattab S, Chavez C, Billingslea-Yoon E, Salazar A, Ellingson BM, Cloughesy TF, Liau LM, Prins RM. TLR agonists polarize interferon responses in conjunction with dendritic cell vaccination in malignant glioma: a randomized phase II Trial. Nat Commun. 2024 May 8;15(1):3882. doi: 10.1038/s41467-024-48073-y. PMID 38719809
- [Derived] Everson RG, Hugo W, Sun L, Antonios J, Lee A, Ding L, Bu M, Khattab S, Chavez C, Billingslea-Yoon E, Salazar A, Ellingson BM, Cloughesy TF, Liau LM, Prins RM. Dendritic Cell Vaccination in Conjunction with a TLR Agonist Polarizes Interferon Immune Responses in Malignant Glioma Patients. Res Sq [Preprint]. 2023 Sep 12:rs.3.rs-3287211. doi: 10.21203/rs.3.rs-3287211/v1. PMID 37790490